CLINICAL TRIAL: NCT05027295
Title: A Randomized Study to Evaluate the Safety and Efficacy of Corneal Collagen Crosslinking Performed With Continuous vs Pulsed UVA Light for Reducing Corneal Curvature in Eyes With Keratoconus and Post-refractive Corneal Ectasia
Brief Title: Accelerated Corneal Collagen Crosslinking for Keratoconus and Ectasia Using Pulse or Continuous UV-A Light
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCEL-CXL-001
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Keratoconus; Corneal Ectasia
Keywords: keratoconus; corneal ectasia; collagen crosslinking; riboflavin; crosslinking; corneal crosslinking
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continuous UVA (Active Comparator): Riboflavin administration one drop every two minutes with administration of 12mW/cm2 of continuous UVA light for 7.5 minute exposure time
  Interventions: Drug: riboflavin ophthalmic solution
- Pulsed UVA (Active Comparator): Riboflavin administration one drop every two minutes with administration of 12mW/cm2 of pulsed UVA light for 15 minute exposure time
  Interventions: Drug: riboflavin ophthalmic solution

INTERVENTIONS:
Drug: riboflavin ophthalmic solution — Administration of riboflavin one drop every 2 minutes during administration of continuous UVA light for 7.5 minutes.
  Arms: Continuous UVA
Drug: riboflavin ophthalmic solution — Administration of riboflavin one drop every 2 minutes during administration of pulsed UVA light for 15 minutes
  Arms: Pulsed UVA

SUMMARY:
Corneal collagen crosslinking has been demonstrated as an effective method of reducing progression of both keratoconus and post-refractive corneal ectasia, as well as decreasing the steepness of the cornea in these pathologies.

Performing an accelerated CXL procedure with pulsed UVA light may increase the oxygenation of the cornea, which may improve the crosslinking efficacy.

DETAILED DESCRIPTION:
This is a prospective, single-site study to analyze the use of continuous vs pulsed UVA light after removal of the epithelium for the collagen crosslinking procedure for keratoconus and post-refractive corneal ectasia. In the standard crosslinking treatment, the cornea is treated with a continuous UVA light treatment with a power of 3mW/cm2 for 30 minutes. CXL treatment can potentially be performed in a shorter period of time by increasing the power of the UVA light and decreasing the exposure time, while maintaining the same total energy delivered to the cornea. This study will compare the efficacy and safety of accelerated crosslinking using either a continuous or pulsed UVA treatment. One group will be randomized to be treated with 12mW/cm2 of continuous UVA light treatment for 7.5 minutes and the other group will be treated with 12mW/cm2 of pulsed UVA light treatment for 15 minutes.

The primary efficacy parameter that will be evaluated over time is maximum keratometry (Kmax) in the randomized eyes for each treatment group. The secondary efficacy parameter is to determine if the two treatment groups are equivalent in their mean Kmax change at 6 months after treatment compared with baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older having a diagnosis of keratoconus or corneal ectasia after corneal refractive surgery
* Presence of central or inferior corneal steepening on the Pentacam map
* Axial topography consistent with keratoconus or post-surgical corneal ectasia
* Contact lens wearers only: removal of contact lenses for the required period of 1 week prior to the screening refraction
* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria:

* Eyes classified as either normal, atypical normal, or keratoconus suspect on the severity grading scheme
* Corneal pachymetry measuring 300 microns or less at the thinnest point measured by Pentacam in the eye(s) to be treated
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:

  1. History of corneal disease (e.g. herpes simplex, herpes zoster keratitis, recurrent corneal erosion syndrome, corneal melt, corneal dystrophy, etc.
  2. Clinically significant scarring in the CXL treatment zone
* A history of chemical injury or delayed healing in the eye(s) to be treated
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests
* Patients with current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Maximum keratometry | 6 months
  The change in maximum keratometry (Kmax) from baseline will be evaluated at 6 months

SECONDARY OUTCOMES:
Mean keratometry | 6 months
  Determine whether the two treatment groups are equivalent in their mean keratometry (meanK) change at 6 months post treatment compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Hersh, MD, Study Director — Cornea and Laser Eye Institute, Hersh Vision Group
Locations (1):
- Cornea and Laser Eye Institute, Hersh Vision Group, Teaneck, New Jersey, United States